CLINICAL TRIAL: NCT02660034
Title: A Phase 1/1b, Open Label, Multiple Dose, Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics and Antitumor Activity of the Anti-PD-1 Monoclonal Antibody BGB-A317 in Combination With the PARP Inhibitor BGB-290 in Subjects With Advanced Solid Tumors
Brief Title: The Safety, Pharmacokinetics and Antitumor Activity of BGB-A317 in Combination With BGB-290 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317/BGB-290_Study_001; 2017-003580-35 (EudraCT Number)
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumors
Keywords: Dose Escalation; Dose Expansion; BGB-A317; BGB-290; Tislelizumab; Pamiparib
MeSH Terms: interventions — tislelizumab; pamiparib

ARMS (2):
- Part A: Dose Escalation Phase (Experimental): Participants received tislelizumab and pamiparib (dose escalation) until determination of the maximum tolerated dose/recommended Phase 2 dose.
  Interventions: Biological: Tislelizumab; Drug: Pamiparib
- Part B: Dose Expansion Phase (Experimental): Participants received tislelizumab and pamiparib (dose expansion).
  Interventions: Biological: Tislelizumab; Drug: Pamiparib

INTERVENTIONS:
Biological: Tislelizumab
  Other Names: BGB-A317
Drug: Pamiparib
  Other Names: BGB-290

SUMMARY:
This trial studied the safety, pharmacokinetics, and antitumor activity of the anti-programmed cell death 1 (PD-1) monoclonal antibody (mAb) BGB-A317 (tislelizumab) in combination with the poly(adenosine diphosphate ribose) polymerase (PARP) inhibitor BGB-290 (pamiparib) in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants voluntarily agreed to participate by giving written informed consent.
2. Must have received standard of care in the primary treatment of their disease.
3. Participants who had the below specified histologically confirmed malignancies that had progressed to the advanced or metastatic stage:

   1. In Part A, the participants must have had an advanced malignancy, including but not limited to high-grade serous cancer of the ovary, fallopian tube, or peritoneum, triple negative breast cancer, small cell lung cancer (SCLC), primary peritoneal cancer, and any tumor likely to harbor DNA damage repair deficiencies susceptible to treatment with a PARP inhibitor or likely to be responsive to a PD-1 blocker.
   2. In Part B, the participants recruited to 1 of the 8 expansion arms must have had advanced solid tumors of the following types:

   Arm 1: Participants with relapsed, platinum-sensitive high-grade epithelial, non-mucinous, ovarian cancer, fallopian tube, or primary peritoneal cancer (EOC) must have met the following criteria:

   i. Must have had at least 2 prior platinum-containing treatments in any treatment setting.

   ii. Must have had platinum-sensitive recurrent disease and must not have progressed (by Response Evaluation Criteria in Solid Tumors [RECIST] v1.1 criteria) within 6 months of the completion of the last platinum-containing line of treatment.

   • Note: Participants may have received additional non-platinum-based chemotherapy for recurrence after prior last platinum-containing regimen if the criteria for platinum sensitivity were met.

   iii. Arm 1a: Participants with relapsed, platinum-sensitive high-grade EOC with either known deleterious or suspected deleterious germline or somatic breast cancer susceptibility gene 1/2 (BRCA1/2) mutations or with homologous recombination deficiency (HRD).

   • If HRD or BRCA1/2 mutation status from archival tissue was unknown or had not been previously evaluated, then the archival tissue must have undergone tissue screening using a validated diagnostic test to determine eligibility. If the diagnostic test result was BRCA1/2 or HRD positive, the participant was eligible for enrollment in Arm 1a.

   iv. Arm 1b: Participants with relapsed, platinum-sensitive high grade EOC who otherwise met the above criteria and were without known germline or somatic BRCA1/2 mutations and without HRD mutation.

   Arm 2: Participants with triple negative breast cancer must have met the following criteria:

   i. 0-1 prior platinum-containing treatment in any treatment setting.

   • Note: participants could have received additional therapy after the last platinum-containing line of treatment if the other eligibility criteria were met.

   ii. Participants who received at least 1 prior treatment but not more than 3 prior lines of treatment in the advanced or metastatic setting.

   iii. Known deleterious or suspected deleterious germline or somatic BRCA1/2 mutations or with documented HRD.

   • If HRD or BRCA1/2 mutation status from archival tissue was unknown or had not been previously evaluated, then the archival tissue must have undergone tissue screening using a validated diagnostic test to determine eligibility. If the diagnostic test result was HRD positive, then the participant was eligible for enrollment in Arm 2.

   • If archival tissue was not available and the participant submitted a fresh tumor biopsy, then the diagnostic test needed to demonstrate somatic BRCA1/2 mutation or HRD positivity.

   Arm 3: Participants with metastatic castration-resistant prostate cancer, including but not limited to mutations in homologous recombination (HR) pathways and/or defined by HRD algorithms, and must have met the following criteria:

   i. May be either chemotherapy-naïve, but must have received prior abiraterone acetate and/or enzalutamide treatment, or have previously had no more than 2 taxane-based chemotherapy lines of treatment, including docetaxel and carbazitaxel. If docetaxel was used more than once, this was considered as 1 line of treatment.

   ii. At least 2 weeks since the completion of prior flutamide, bicalutamide, and nilutimide, or enzalutamide and abiraterone treatment.

   iii. Documented prostate cancer with one of the following:
   * Surgically or medically castrated. The testosterone levels did not need to be checked if the participant had undergone surgical castration for > 4 months. Participants receiving chemical castration should have had testosterone levels checked at baseline and confirmed to be in the castrate levels (< 0.5 ng/mL or 1.735 nM). In all cases, the luteinizing hormone-releasing hormone antagonist/agonist was to be continued in these participants.
   * Participants with only non-measurable bone lesions must have had disease progression based on Prostate Cancer Clinical Trials Working Group with 2 or more new lesions or have had prostate-specific antigen progression before enrolment.

   iv. Known deleterious or suspected deleterious germline or somatic BRCA1/2 mutations or with documented HRD.
   * If HRD or BRCA1/2 mutation status from archival tissue was unknown or had not been previously evaluated, then the archival tissue must have undergone tissue screening using a validated diagnostic test to determine eligibility. If the diagnostic test result was HRD positive, then the participant was be eligible for enrollment in Arm 3.
   * If archival tissue was not available and the participant summitted a fresh tumor biopsy, then the diagnostic test needed to demonstrate somatic BRCA1/2 mutation or HRD positivity.

   Arm 4: Participants with extensive-stage disease SCLC must have met the following criteria:

   i. Received at least 1 and not more than 2 prior lines of treatment; ii. At least 1 prior line of treatment must have contained a platinum agent

   Arm 5: Participants with human epidermal growth factor receptor-2 (HER2)-negative gastric or gastroesophageal junction cancer must have met the following criteria:

   i. May have received at least 1 and not more than 2 prior lines of treatment

   Arm 6: Participants with locally advanced or metastatic urothelial (muscle-invasive bladder, ureter, urethra, or renal pelvis) cancer must have met the following criteria:

   i. Received at least 1 and not more than 2 prior lines of treatment in the advanced or metastatic disease setting; ii. At least 1 prior line of treatment must have contained a platinum agent

   Arm 7: Participants with advanced or metastatic pancreatic adenocarcinoma must have met the following criteria:

   i. Received at least 1 but not more than 2 lines of treatment in either an advanced or metastatic setting; ii. At least 1 prior treatment for advanced or metastatic disease must have contained a platinum agent; iii. Participants with known deleterious germline or somatic BRCA1/2 mutation could be considered for the study even if platinum naïve.

   Arm 8: (Note: Closed to enrollment) Participants with advanced or metastatic recurrent non-ovarian gynecological cancers (endometrial cancer, cancer of the cervix and participants with tumors known to be mismatch repair deficient or HRD positive) must have met the following criteria:

   i. Participants with a complete response, partial response, or stable disease from at least 1 prior platinum-containing treatment in any treatment setting; ii. The Sponsor medical monitor would approve tumor types for Arm 8 prior to screening.

   • Note: Excluded tumor types included participants with bone or soft tissue sarcoma; central nervous system (CNS) malignancies; colorectal cancer (except microsatellite instability-high colorectal cancer is permitted); cutaneous or ocular melanoma; hematologic malignancies; HER2-negative breast cancer without BRCA mutation; mesothelioma, papillary, follicular, medullary or Hürthle cell thyroid cancer; unknown primary malignancy.
4. Participants who were treated with chemotherapy or any investigational therapies, if eligible, must have completed at least 4 weeks or at least 5 half-lives (whichever is longer, but no less than 3 weeks) before the study drug administration, and all adverse events (AEs) had either returned to baseline or stabilized.
5. At least 2 weeks from palliative radiotherapy.
6. Participants must have had archival tumor tissue or agree to a tumor biopsy for mutation and biomarkers analysis unless previously discussed with Sponsor's medical monitor or its designee (fresh tumor biopsies were recommended at baseline in participants with readily accessible tumor lesions and who consented to the biopsies). Participants with ovarian, fallopian tube, primary peritoneal, or breast cancer in Part A and all participants enrolled in Part B must also have agreed to provide fresh blood sample at the baseline for the evaluation of BRCA mutations and/or confirmation of prior BRCA results or other HR deficiency mutations, even if it was previously tested.
7. Participants must have had measurable disease as defined in RECIST v1.1. Participants with metastatic castration-resistant prostate cancer and epithelial, non-mucinous, ovarian cancer, fallopian tube, or primary peritoneal cancer may have used separate disease-specific criteria.
8. Male or female ≥ 18 years of age on the day of signing informed consent.
9. Must have had an Eastern Cooperative Oncology Group Performance Status ≤ 1.
10. Must have had a life expectancy ≥ 12 weeks.
11. Must have had adequate organ function.
12. Females of childbearing potential must have been willing to use a highly effective method of birth control for the duration of the study, and for at least 6 months after the last dose of investigational drug, and have had a negative serum pregnancy test within 7 days of the first dose of study drug(s).
13. Non-sterile males and their female partners must have been willing to use a highly effective method of birth control for the duration of the study and for at least 6 months after the last dose of investigational drug. Nonsterile males must have avoided sperm donation for the duration of the study and for at least 6 months after last study drug.
14. Females must have agreed not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study drug administration.

Key Exclusion Criteria:

1. Participants with ovarian cancer who have platinum-resistant/refractory disease, defined as progressive disease at the first tumor assessment while receiving platinum-containing chemotherapy.
2. Participant had history of severe hypersensitivity reactions to other mAbs.
3. Any major surgery within 28 days before first dose of study drugs.
4. Prior allogeneic stem cell transplantation or organ transplantation.
5. Participants with toxicities (as a result of prior anticancer therapy) that had not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (for example, alopecia, neuropathy and specific laboratory abnormalities).
6. Concurrent participation in another clinical trial.
7. Prior malignancy within the previous 2 years except for locally curable non-melanoma dermatologic cancers that had been apparently cured, such as basal or squamous cell skin cancer, or carcinoma in situ of the skin, cervix, breast, bladder, or prostate.
8. Symptomatic CNS metastasis or leptomeningeal disease. Note: Baseline magnetic resonance imaging of the brain and spinal cord was required for SCLC participants enrolled in Arm 4 if they had a history of CNS disease.

   Note: Participants with previously treated CNS metastatic disease were eligible for any arm if CNS metastatic disease was asymptomatic, clinically stable, and did not require corticosteroids or anticonvulsants within a minimum of 4 weeks of enrollment.
9. Prior therapies targeting PD-1, programmed death-ligand 1 (PD-L1), or PARP.
10. Active autoimmune diseases or history of autoimmune diseases that may have relapsed.

    Note: Participants with the following diseases were not excluded and may have proceeded to further screening:
    1. Controlled Type I diabetes;
    2. Hypothyroidism managed with no treatment other than with hormone replacement therapy;
    3. Controlled celiac disease;
    4. Skin diseases not requiring systemic treatment (for example, vitiligo, psoriasis, alopecia);
    5. Any other disease that was not expected to recur in the absence of external triggering factors.
11. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication within 2 weeks of the study drug administration.

    Note: Participants who were currently or had previously been on any of the following steroid regimens were not excluded:
    1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent);
    2. Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption;
    3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (for example, for contrast dye allergy) or for the treatment of a non-autoimmune condition (for example, delayed-type hypersensitivity reaction caused by contact allergen).
12. With severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, et cetera.
13. History of interstitial lung disease, non-infectious pneumonitis or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung diseases, et cetera.
14. History of non-viral hepatitis or cirrhosis.
15. Positive human immunodeficiency virus status.
16. A known history of hepatitis B virus or hepatitis C virus infection.
17. History of alcohol abuse.
18. Underlying medical conditions or alcohol or drug abuse or dependence that, in the investigator's opinion, would be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs; or insufficient compliance during the study according to investigator's judgement.
19. Inability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening, or otherwise altering the product formulation. Participants should not have had gastrointestinal illnesses that would have precluded the absorption of pamiparib, which was an oral agent.
20. Had been administered a live vaccine within 4 weeks (28 days) of initiation of study therapy.
21. Any of the following cardiovascular criteria:

    1. Current evidence of cardiac ischemia;
    2. Current symptomatic pulmonary embolism;
    3. Acute myocardial infarction ≤ 6 months prior to Day 1;
    4. Heart failure of New York Heart Association Classification III or IV ≤ 6 months prior to Day 1;
    5. Grade ≥ 2 ventricular arrhythmia ≤ 6 months prior to Day 1;
    6. History of cerebrovascular accident within 6 months before first dose of study drugs.
22. Use or had anticipated need for food or drugs known to be strong or moderate cytochrome P450 (CYP)3A inhibitors or strong CYP3A inducers ≤ 10 days (or ≤ 5 half-lives, whichever is shorter) prior to Day 1.

Note: Other protocol-defined Inclusion/Exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (29):
- United States (12):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Texas Oncology, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (10):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Mid North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Westmead Hospital, Parramatta, New South Wales
  - Prince of Wales, Randwick, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Icon Cancer Care, Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- France (2):
  - Institut Gustave Roussy, Paris
  - Centre Eugene Marquis, Rennes
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Capital and Coast District Health Board, Wellington
- Spain (2):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia
- Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Friedlander M, Meniawy T, Markman B, Mileshkin L, Harnett P, Millward M, Lundy J, Freimund A, Norris C, Mu S, Wu J, Paton V, Gao B. Pamiparib in combination with tislelizumab in patients with advanced solid tumours: results from the dose-escalation stage of a multicentre, open-label, phase 1a/b trial. Lancet Oncol. 2019 Sep;20(9):1306-1315. doi: 10.1016/S1470-2045(19)30396-1. Epub 2019 Aug 1. PMID 31378459
- [Derived] Friedlander M, Mileshkin L, Lombard J, Frentzas S, Gao B, Wilson M, Meniawy T, Baron-Hay S, Briscoe K, McCarthy N, Fountzilas C, Cervantes A, Ge R, Wu J, Spira A. Pamiparib in combination with tislelizumab in patients with advanced solid tumours: results from the dose-expansion stage of a multicentre, open-label, phase I trial. Br J Cancer. 2023 Sep;129(5):797-810. doi: 10.1038/s41416-023-02349-0. Epub 2023 Jul 20. PMID 37474720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A: A total of 49 participants with advanced solid tumors were enrolled in Part A of the study (dose escalation phase) at a total of 5 sites or community oncology centers in Australia. Part B: A total of 180 participants with advanced solid tumors were enrolled in Part B of the study (dose expansion phase).
Groups:
- Part A: Dose Escalation Phase - Cohort 1: Participants received tislelizumab (2 milligrams/kilogram [mg/kg] once every 3 weeks [Q3W] intravenously [IV]) with pamiparib (20 mg twice daily) (dose escalation) until determination of the maximum tolerated dose/recommended Phase 2 dose (MTD/RP2D).
- Part A: Dose Escalation Phase - Cohort 2: Participants received tislelizumab (2 mg/kg Q3W IV) with pamiparib (40 mg twice daily) (dose escalation) until determination of the MTD/RP2D.
- Part A: Dose Escalation Phase - Cohort 3: Participants received tislelizumab (2 mg/kg Q3W IV) with pamiparib (60 mg twice daily) (dose escalation) until determination of the MTD/RP2D.
- Part A: Dose Escalation Phase - Cohort 4: Participants received tislelizumab (200 mg/kg Q3W IV) with pamiparib (40 mg twice daily) (dose escalation) until determination of the MTD/RP2D.
- Part A: Dose Escalation Phase - Cohort 5: Participants received tislelizumab (200 mg/kg Q3W IV) with pamiparib (60 mg twice daily) (dose escalation) until determination of the MTD/RP2D.
- Part B: Dose Expansion Phase - Arm 1a: Participants with relapsed, platinum-sensitive, high-grade epithelial, non-mucinous, ovarian cancer, fallopian tube, or primary peritoneal cancer (EOC) with either known germline or somatic breast cancer susceptibility gene 1/2 (BRCA1/2) mutations or with homologous recombination deficiency (HRD) received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily.
- Part B: Dose Expansion Phase - Arm 1b: Participants with relapsed, platinum-sensitive, high-grade EOC without either known germline or somatic BRCA1/2 mutations and without known HRD received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. Participants must have received at least 2 prior lines of platinum-containing chemotherapy.
- Part B: Dose Expansion Phase - Arm 2: Participants with triple negative breast cancer (TNBC) with either known germline or somatic BRCA1/2 mutations or with documented HRD received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. Participants could have been treated with at least 1 but no more than 3 prior lines of treatment.
- Part B: Dose Expansion Phase - Arm 3: Participants with metastatic castration-resistant prostate cancer (mCRPC) with either known germline or somatic BRCA1/2 mutations or with documented HRD received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. Chemotherapy-naïve participants must have received prior abiraterone acetate or enzalutamide treatment.
- Part B: Dose Expansion Phase - Arm 4: Participants with extensive-stage disease small cell lung cancer (SCLC) treated with at least 1 but no more than 2 prior lines of treatment, at least 1 must have included a platinum agent, received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily.
- Part B: Dose Expansion Phase - Arm 5: Participants with human epidermal growth factor receptor-2 (HER2)-negative gastric or gastroesophageal junction cancer received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. Participants with HER2-negative disease could be treated with at least 1 but no more than 2 prior lines of treatment.
- Part B: Dose Expansion Phase - Arm 6: Participants with locally advanced or metastatic urothelial (muscle invasive bladder, ureter, urethra, or renal pelvis) cancer treated with at least 1 but no more than 2 prior lines of treatment, including a prior platinum-containing chemotherapy, received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily.
- Part B: Dose Expansion Phase - Arm 7: Participants with advanced or metastatic pancreatic adenocarcinoma treated with at least 1 but no more than 2 prior lines of therapy received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. At least 1 prior treatment for advanced or metastatic disease must have contained a platinum agent. Any potential participant with a known deleterious germline or somatic BRCA was eligible even if platinum naïve.
- Part B: Dose Expansion Phase - Arm 8: Participants who were expected to benefit from the combination of a poly (ADP-ribose) polymerase (PARP) inhibitor and a programmed cell death 1 (PD-1) inhibitor received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. This arm included participants with recurrent non-ovarian gynecological cancers (endometrial cancer, cancer of the cervix, and participants with tumors known to be mismatch repair [MMR] deficient or HRD positive) that were not eligible for inclusion in any other arms of the study. This was an exploratory signal seeking arm.
Period: Overall Study
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5 | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Started | 12 | 12 | 6 | 13 | 6 | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
Received At Least 1 Dose of Study Drug(s) (Safety Analysis Set) | 12 | 12 | 6 | 13 | 6 | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 12 | 6 | 13 | 6 | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
Not completed — Progressive Disease (Radiographic) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease (Clinical) | 7 | 8 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Participant moved into special access scheme | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 13 | 14 | 10 | 9 | 21 | 17 | 15 | 18 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participants transferred to LTE | 0 | 0 | 0 | 0 | 0 | 10 | 8 | 8 | 10 | 1 | 2 | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of tislelizumab and/or pamiparib.
Groups:
- Part A: Dose Escalation Phase - Cohort 1: Participants received tislelizumab (2 mg/kg Q3W IV) with pamiparib (20 mg twice daily) (dose escalation) until determination of the MTD/RP2D.
- Part B: Dose Expansion Phase - Arm 1a: Participants with relapsed, platinum-sensitive, high-grade EOC with either known BRCA1/2 mutations or with HRD received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily.
- Part B: Dose Expansion Phase - Arm 2: Participants with TNBC with either known germline or somatic BRCA1/2 mutations or with documented HRD received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. Participants could have been treated with at least 1 but no more than 3 prior lines of treatment.
- Part B: Dose Expansion Phase - Arm 3: Participants with mCRPC with either known germline or somatic BRCA1/2 mutations or with documented HRD received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. Chemotherapy-naïve participants must have received prior abiraterone acetate or enzalutamide treatment.
- Part B: Dose Expansion Phase - Arm 4: Participants with extensive-stage disease SCLC treated with at least 1 but no more than 2 prior lines of treatment, at least 1 must have included a platinum agent, received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily.
- Part B: Dose Expansion Phase - Arm 5: Participants with HER2-negative gastric or gastroesophageal junction cancer received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. Participants with HER2-negative disease could be treated with at least 1 but no more than 2 prior lines of treatment.
- Part B: Dose Expansion Phase - Arm 8: Participants who were expected to benefit from the combination of a PARP inhibitor and a PD-1 inhibitor received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. This arm included participants with recurrent non-ovarian gynecological cancers (endometrial cancer, cancer of the cervix, and participants with tumors known to be MMR deficient or HRD positive) that were not eligible for inclusion in any other arms of the study. This was an exploratory signal seeking arm.
- Total: Total of all reporting groups
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5 | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8 | Total
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6 | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.39) | 58.6 (9.52) | 54.5 (11.27) | 61.8 (11.42) | 64.3 (5.96) | 59.5 (10.71) | 69.1 (8.68) | 50.4 (12.41) | 68.0 (8.89) | 64.2 (9.87) | 58.5 (13.71) | 68.9 (10.45) | 63.3 (9.11) | 60.1 (16.20) | 62.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 5 | 12 | 5 | 23 | 23 | 19 | 0 | 10 | 3 | 6 | 9 | 5 | 140
  Male | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 20 | 13 | 17 | 15 | 12 | 5 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 7
  Not Hispanic or Latino | 12 | 12 | 6 | 13 | 6 | 22 | 22 | 16 | 18 | 21 | 17 | 17 | 19 | 9 | 210
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 2 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
  White | 10 | 12 | 5 | 11 | 6 | 20 | 23 | 17 | 18 | 18 | 16 | 18 | 19 | 8 | 201
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 3 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number Of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not. All AEs reported are treatment-emergent, which was defined as having a reported onset time or worsening in severity on or after the date of the first dose of study treatment through 30 days after the last dose (permanent discontinuation of study treatment) or initiation of new anticancer therapy. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: From Day 1 up to 4 years and 7 months
Population: The safety analysis set (SAF) included all participants (both parts) who received at least one dose of tislelizumab and/or pamiparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
Participants | 12 | 12 | 6 | 13 | 6

2. Primary Outcome: Part A: Number Of Participants Experiencing Dose-limiting Toxicity (DLT)
Description: DLT was defined as an AE or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications, and occurs during the first 21 days following the first dose of tislelizumab and pamiparib in Cycle 1 and meets protocol-specified criteria. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: 21 days following the first dose of tislelizumab and pamiparib in Cycle 1
Population: SAF included all participants (both parts) who received at least one dose of tislelizumab and/or pamiparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
Participants | 0 | 0 | 0 | 2 | 2

3. Primary Outcome: Part B: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) and partial response (PR).
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Dose Expansion Phase - Arm 1a: Participants with relapsed, platinum-sensitive, high-grade EOC with either known germline or somatic BRCA1/2 mutations or with HRD received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily.
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
Participants | 7 | 3 | 9 | 4 | 2 | 2 | 6 | 0 | 3

4. Primary Outcome: Part B: Progression-free Survival (PFS)
Description: PFS was defined as the time from first dose of study medication to the first documented objective disease progression or death due to any cause, whichever occurred first.
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 7
month | 8.2 [5.2 to 11.8] | 3.5 [1.9 to 7.6] | 8.4 [3.9 to 19.0] | 10.4 [4.3 to 16.2] | 2.0 [1.7 to 2.3] | 2.1 [1.9 to 4.1] | 3.5 [1.9 to 7.5] | 1.9 [1.1 to 2.1] | 2.2 [1.2 to 24.4]

5. Primary Outcome: Part B: Duration Of Response (DOR)
Description: DOR, defined as the time from the first determination of an objective response, was assessed by investigator per Response Evaluation Criteria in Solid Tumors v1.1 until the first documentation of progression or death, whichever occurred first. Results are reported only for arms with responders.
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 7 | 3 | 9 | 4 | 2 | 2 | 6 | 3
months | 11.2 [6.2 to NA] — NA = not estimable due to insufficient number of participants with events | 6.2 [3.8 to NA] — NA = not estimable due to insufficient number of participants with events | 17.1 [3.0 to NA] — NA = not estimable due to insufficient number of participants with events | NA [4.1 to NA] — NA = not estimable due to insufficient number of participants with events | 6.2 [4.3 to 8.1] | NA [NA to NA] — NA = not estimable due to insufficient number of participants with events | NA [5.7 to NA] — NA = not estimable due to insufficient number of participants with events | NA [22.4 to NA] — NA = not estimable due to insufficient number of participants with events

6. Primary Outcome: Part B: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a best overall response of CR, PR, and stable disease (SD).
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
Participants | 21 | 11 | 14 | 15 | 7 | 7 | 12 | 2 | 4

7. Primary Outcome: Part B: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with a best overall response of CR, PR, and SD lasting ≥ 24 weeks.
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
Participants | 15 | 7 | 11 | 10 | 4 | 4 | 8 | 1 | 3

8. Primary Outcome: Part B: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study drug to death due to any cause.
Time Frame: From Day 1 Every 3 months following completion or discontinuation of the treatment (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
month | 20.9 [13.5 to NA] — NA = not estimable due to insufficient number of participants with events | 18.7 [6.1 to 27.0] | 15.8 [10.4 to NA] — NA =not estimable due to insufficient number of participants with events | 21.2 [10.5 to NA] — NA = not estimable due to insufficient number of participants with events | 6.9 [3.3 to 11.5] | 7.4 [3.3 to 13.4] | 8.4 [4.4 to 17.1] | 4.1 [2.9 to 5.0] | 4.1 [1.2 to 19.5]

9. Secondary Outcome: Part A: Minimum Observed Plasma Concentration (Ctrough) Of Tislelizumab
Time Frame: Cycle 4 Day 1 (0 hours and 4 hours) post dose
Population: The PK Analysis Set included participants in the Safety Analysis Set for whom at least one PK parameter can be derived for either pamiparib or tislelizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 5 | 8 | 4 | 7 | 2
nanogram/milliliter
  Cycle 4 Day 1 (Pre-dose) | 23530 (48.02) | 26040 (58.04) | 26160 (23.69) | 30330 (58.28) | 53700 (81.62)
  Cycle 4 Day 1 (4 h) | 74260 (20.70) | 66250 (47.28) | 69020 (16.47) | 104300 (35.31) | 119600 (33.83)

10. Secondary Outcome: Part A: Ctrough Of Pamiparib
Time Frame: Cycle 2 Day 1 (Pre-dose and 7 hours Post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
nanogram/milliliter
  Cycle 2 Day 1 (Pre-dose): number analyzed (Participants) | 10 | 11 | 5 | 9 | 4
  Cycle 2 Day 1 (Pre-dose) | 772.9 (164.6) | 1258 (62.13) | 1209 (42.18) | 1876 (60.41) | 2754 (48.69)
  Cycle 2 Day 1 (7 h): number analyzed (Participants) | 9 | 11 | 5 | 11 | 4
  Cycle 2 Day 1 (7 h) | 824.8 (130.6) | 1469 (38.14) | 1717 (55.56) | 2070 (47.36) | 2969 (48.77)

11. Secondary Outcome: Part A: Maximum Observed Plasma Concentration At Steady State (Cmax,ss) Of Pamiparib
Time Frame: Cycle 2 Day 1 (Pre-dose and 7 hours Post-dose)
Population: as for outcome 9
Measure: Number; unit: nanogram/milliliter
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
nanogram/milliliter | 1457 | 2497 | 2985 | 2586 | 3189

12. Secondary Outcome: Part A: Time To Reach Maximum Plasma Concentration At Steady State (Tmax,ss) Of Pamiparib
Time Frame: Cycle 2 Day 1 (Pre-dose and 7 hours Post-dose)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: hour
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
hour | 1.0 [0.60 to 6.2] | 1.1 [0.42 to 4.0] | 1.0 [1.0 to 7.1] | 1.9 [0.45 to 7.0] | 2.0 [0.92 to 3.8]

13. Secondary Outcome: Part A: Ctrough At Steady State (Ctrough,ss) Of Pamiparib
Time Frame: Cycle 2 Day 1 (Pre-dose and 7 hours Post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
nanogram/milliliter | 494 (130) | 1170 (66) | 1151 (97) | 2135 (39) | 2554 (2.5)

14. Secondary Outcome: Part A: ORR
Description: ORR was defined as the percentage of participants with a best overall response of CR and PR.
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: EFF included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
Participants | 1 | 3 | 0 | 3 | 3

15. Secondary Outcome: Part A: PFS
Description: as for outcome 4
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: EFF included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
Days | 64 [46 to 125] | 77 [42 to 568] | 190 [39 to 963] | 107 [58 to 249] | 373 [106 to 516]

16. Secondary Outcome: Part A: DCR
Description: DCR was defined as the percentage of participants with a best overall response of CR, PR, and SD.
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
Participants | 3 | 6 | 5 | 7 | 5

17. Secondary Outcome: Part A: CBR
Description: CBR was defined as the percentage of participants with a best overall response of CR, PR, and SD lasting ≥ 24 weeks.
Time Frame: Starting from Day 1 until disease progression (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Median (Standard Deviation); unit: week
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
week | 2 (16.7) | 5 (41.7) | 4 (66.7) | 4 (30.8) | 4 (66.7)

18. Secondary Outcome: Part A: OS
Description: OS was defined as the time from the date of first dose of study drug to death due to any cause.
Time Frame: Starting from Day 1 Every 3 months following completion or discontinuation of the treatment (up to 4 years and 7 months)
Population: The efficacy evaluable set (EFF) included participants in the SAF who had measurable or evaluable disease at baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
Days | 259 [46 to 437] | 413 [54 to 1127] | NA [107 to NA] — NA = Not estimable due to insufficient number of participants with events | 434 [128 to 577] | NA [178 to NA] — NA = Not estimable due to insufficient number of participants with events

19. Secondary Outcome: Part A: Percentage Of Participants With Anti-drug Antibodies (ADAs) For Tislelizumab
Description: Immunogenicity was summarized by participants who were ADA positive and developed detectable ADAs.
Time Frame: Within 24 hours before the start of the first dose of tislelizumab in Cycle 1, Day 8 of Cycle 1, and Day 1 of Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 9, and Cycle 17
Population: The Antidrug Antibody (ADA) Analysis Set included participants who received ≥ 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5
Number analyzed (Participants) | 12 | 12 | 6 | 13 | 6
Participants | 3 | 1 | 0 | 1 | 0

20. Secondary Outcome: Part B: Number Of Participants Experiencing AEs
Description: as for outcome 1
Time Frame: Day 1 of Cycle 1 up to 4 years and 7 months
Population: SAF will include all participants (both parts) who received at least one dose of tislelizumab and/or pamiparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 10
Participants | 23 | 23 | 19 | 20 | 23 | 20 | 21 | 21 | 9

21. Secondary Outcome: Part B: Ctrough Of Tislelizumab
Description: As pre-specified in the protocol, pharmacokinetic evaluations were performed for all Part B dose expansion arms combined.
Time Frame: Cycle 4 Day 1 ( 0 hours and 4 hours post dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Groups:
- Part B: Dose Expansion Phase: Participants received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily.
Arm/Group | Part B: Dose Expansion Phase
Number analyzed (Participants) | 180
nanogram/milliliter | 46060 (36)

22. Secondary Outcome: Part B: Maximum Observed Plasma Concentration (Cmax) Of Tislelizumab
Description: as for outcome 21
Time Frame: Cycle 4 Day 1 ( 0 hours and 4 hours) post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Part B: Dose Expansion Phase
Number analyzed (Participants) | 180
nanogram/milliliter | 99408 (20)

23. Secondary Outcome: Part B: Ctrough Of Pamiparib
Description: as for outcome 21
Time Frame: Cycle 2 Day 1 (7 hours Post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Part B: Dose Expansion Phase
Number analyzed (Participants) | 180
nanogram/milliliter | 1161 (80)

24. Secondary Outcome: Part B: Cmax Of Pamiparib
Description: as for outcome 21
Time Frame: Cycle 2 (7 hours Post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Part B: Dose Expansion Phase
Number analyzed (Participants) | 180
nanogram/milliliter | 1850 (63)

25. Secondary Outcome: Part B: Percentage Of Participants With ADAs For Tislelizumab
Description: Immunogenicity was summarized by participants who developed detectable ADAs. Treatment-emergent ADAs: sum of both treatment-induced ADAs and treatment-boosted ADAs.
Time Frame: 24 hours predose of Day 1 of every cycle
Population: The Antidrug Antibody (ADA) Analysis Set included participants who received ≥ 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
Number analyzed (Participants) | 19 | 18 | 16 | 18 | 21 | 19 | 19 | 17 | 9
Participants
  Treatment-emergent ADA | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-induced ADA | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
  Persistent ADA Response | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Transient ADA Response | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  NAb Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through 4 years and 7 months
Groups:
- Part B: Dose Expansion Phase - Arm 7: Participants with advanced or metastatic pancreatic adenocarcinoma treated with at least 1 but no more than 2 prior lines of therapy received tislelizumab 200 mg IV Q3W + pamiparib 40 mg orally twice daily. At least 1 prior treatment for advanced or metastatic disease must have contained a platinum agent. Any potential participant with a known deleterious germline or somatic BRCA was eligible even if platinum-naïve.
Arm/Group | Part A: Dose Escalation Phase - Cohort 1 | Part A: Dose Escalation Phase - Cohort 2 | Part A: Dose Escalation Phase - Cohort 3 | Part A: Dose Escalation Phase - Cohort 4 | Part A: Dose Escalation Phase - Cohort 5 | Part B: Dose Expansion Phase - Arm 1a | Part B: Dose Expansion Phase - Arm 1b | Part B: Dose Expansion Phase - Arm 2 | Part B: Dose Expansion Phase - Arm 3 | Part B: Dose Expansion Phase - Arm 4 | Part B: Dose Expansion Phase - Arm 5 | Part B: Dose Expansion Phase - Arm 6 | Part B: Dose Expansion Phase - Arm 7 | Part B: Dose Expansion Phase - Arm 8
All-Cause Mortality (participants affected / at risk) | 11/12 | 9/12 | 2/6 | 10/13 | 3/6 | 13/23 | 14/23 | 10/19 | 9/20 | 21/23 | 17/20 | 15/21 | 20/21 | 8/10
Serious Adverse Events (participants affected / at risk) | 5/12 | 5/12 | 3/6 | 6/13 | 5/6 | 6/23 | 16/23 | 7/19 | 8/20 | 14/23 | 10/20 | 13/21 | 8/21 | 8/10
Other Adverse Events (participants affected / at risk) | 12/12 | 11/12 | 5/6 | 12/13 | 6/6 | 21/23 | 22/23 | 16/19 | 13/20 | 15/23 | 17/20 | 14/21 | 18/21 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Part A: Dose Escalation Phase - Cohort 1 (N=12) | Part A: Dose Escalation Phase - Cohort 2 (N=12) | Part A: Dose Escalation Phase - Cohort 3 (N=6) | Part A: Dose Escalation Phase - Cohort 4 (N=13) | Part A: Dose Escalation Phase - Cohort 5 (N=6) | Part B: Dose Expansion Phase - Arm 1a (N=23) | Part B: Dose Expansion Phase - Arm 1b (N=23) | Part B: Dose Expansion Phase - Arm 2 (N=19) | Part B: Dose Expansion Phase - Arm 3 (N=20) | Part B: Dose Expansion Phase - Arm 4 (N=23) | Part B: Dose Expansion Phase - Arm 5 (N=20) | Part B: Dose Expansion Phase - Arm 6 (N=21) | Part B: Dose Expansion Phase - Arm 7 (N=21) | Part B: Dose Expansion Phase - Arm 8 (N=10)
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Pyoderma streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/9 | 0/11 | 0/5 | 1/12 | 0/5 | 0 | 0 | 0 | 0/0 | 0/10 | 0/3 | 0/6 | 0/9 | 0/5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Part A: Dose Escalation Phase - Cohort 1 (N=12) | Part A: Dose Escalation Phase - Cohort 2 (N=12) | Part A: Dose Escalation Phase - Cohort 3 (N=6) | Part A: Dose Escalation Phase - Cohort 4 (N=13) | Part A: Dose Escalation Phase - Cohort 5 (N=6) | Part B: Dose Expansion Phase - Arm 1a (N=23) | Part B: Dose Expansion Phase - Arm 1b (N=23) | Part B: Dose Expansion Phase - Arm 2 (N=19) | Part B: Dose Expansion Phase - Arm 3 (N=20) | Part B: Dose Expansion Phase - Arm 4 (N=23) | Part B: Dose Expansion Phase - Arm 5 (N=20) | Part B: Dose Expansion Phase - Arm 6 (N=21) | Part B: Dose Expansion Phase - Arm 7 (N=21) | Part B: Dose Expansion Phase - Arm 8 (N=10)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 1 | 3 | 5 | 3 | 1 | 0 | 4 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 1 | 1 | 1 | 4 | 8 | 5 | 6 | 3 | 8 | 3 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 4 | 5 | 3 | 10 | 6 | 8 | 4 | 4 | 6 | 6 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 4 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 10 | 4 | 10 | 5 | 18 | 17 | 15 | 8 | 8 | 7 | 12 | 12 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 7 | 1 | 5 | 3 | 6 | 5 | 8 | 3 | 2 | 4 | 4 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 7 | 3 | 7 | 4 | 10 | 15 | 12 | 12 | 5 | 11 | 9 | 9 | 5
Influenza like illness (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 2 | 2 | 0 | 1 | 3 | 1 | 2 | 1 | 0 | 2 | 2 | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 2 | 2 | 1 | 5 | 1 | 7 | 3 | 2 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 3 | 2 | 4 | 3 | 1 | 3 | 1 | 3 | 4 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0/9 | 1/11 | 2/5 | 0/12 | 0/5 | 0 | 0 | 0 | 0/0 | 0/10 | 0/3 | 0/6 | 0/9 | 0/5
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 3 | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 1 | 2 | 1 | 0 | 3 | 6 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 1 | 5 | 3 | 3 | 5 | 1 | 1 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 0 | 3 | 8 | 3 | 5 | 5 | 5 | 4 | 3 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 3 | 6 | 4 | 1 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 2 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 5 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 3 | 3 | 0 | 1 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 1 | 3 | 2 | 4 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 2 | 2 | 1 | 5 | 3 | 5 | 3 | 3 | 3 | 2 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 0 | 3 | 1 | 1 | 1 | 5 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 4 | 1 | 1 | 1 | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 4 | 3 | 5 | 2 | 10 | 5 | 3 | 2 | 5 | 5 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1 | 1 | 1 | 3 | 5 | 3 | 6 | 2 | 1 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 3 | 2 | 4 | 0 | 3 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 2 | 2 | 8 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 2 | 2 | 9 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 3 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 6 | 4 | 2 | 2 | 8 | 3 | 3 | 5 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 4 | 0 | 0 | 2 | 2 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 1 | 2 | 4 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 5 | 0 | 2 | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 2 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 3 | 2 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 3 | 0 | 3 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/9 | 0/11 | 0/5 | 1/12 | 0/5 | 0 | 0 | 0 | 0/0 | 0/10 | 0/3 | 0/6 | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT02660034/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT02660034/SAP_001.pdf